CLINICAL TRIAL: NCT07355920
Title: Clinical Evaluation of Alkasite Composite as a Final Restoration for Pulpotomized Primary Molars.
Brief Title: Use of Alkasite for Postpulpotomy Restoration
Acronym: Cention-Forte
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Manar Taha Mokhtar Hamed Elsayed, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #P-PED-6-24-2204
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Dentistry; Post Pulpotomy Restoration
Keywords: cention forte; tetric n ceram; alkasite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: Study group :Alkasite( cention forte ) (Experimental): 25 primary molars were restored with an Alkasite composite Cention-forte after Formocresol pulpotomy.
  Interventions: Procedure: Cention Forte
- Group II :Control group: Tetric N-Ceram (Active Comparator): 25 primary molars were restored with Tetric® N-Ceram bulk-fill composite after Formocresol pulpotomy.
  Interventions: Procedure: Tetric® N-Ceram

INTERVENTIONS:
Procedure: Cention Forte — 25 primary molars were restored with an Alkasite composite Cention-forte after Formocresol pulpotomy.
  Other Names: alkasite
  Arms: Group I: Study group :Alkasite( cention forte )
Procedure: Tetric® N-Ceram — 5 primary molars were restored with Tetric® N-Ceram bulk-fill composite after Formocresol pulpotomy.
  Other Names: bulk-fill composite
  Arms: Group II :Control group: Tetric N-Ceram

SUMMARY:
The aim of this study will be directed to:

Evaluate the clinical performance of alkasite composite as a final restoration for pulpotomized primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Deep carious vital primary molars at site 1, 2, and size 3 according to the SI/STA classification of caries.
* Healthy children free from systemic diseases.
* Cooperative patient: Frankel rating 3,4.

Radiographically:

* Deep caries approximating the pulp.
* Roots with no more than one-third physiologic resorption.
* Normal lamina dura and periodontal ligament space.

Exclusion Criteria:

* Patients with bruxism.
* Clinical signs or symptoms of irreversible pulpitis or pulp degeneration.
* Parents refuse treatment.

Radiographically:

* Furcation involvement.
* periapical lesion.
* Pathologic resorption (internal or external).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of the final restoration according to USPHS Criteria | at 3, 6, and 9 months
  Clinical evaluation of the final restoration is done according to the modified united states public health service USPHS Criteria for direct clinical evaluation of restoration

CONTACTS AND LOCATIONS:
Overall Officials: Faten Abu Taleb, Study Chair — faculty of dentistry Tanta university
Locations (1):
- The clinical study was carried out at the clinic of Pediatric and Preventive Dentistry Department, Faculty of dentistry, Tanta university., Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur K, Suneja B, Jodhka S, Saini RS, Chaturvedi S, Bavabeedu SS, Alhamoudi FH, Cicciu M, Minervini G. Comparison between Restorative Materials for Pulpotomised Deciduous Molars: A Randomized Clinical Study. Children (Basel). 2023 Feb 1;10(2):284. doi: 10.3390/children10020284. PMID 36832414